CLINICAL TRIAL: NCT05489939
Title: Safety and Efficacy of Compound Methyl Salicylate Liniment for Topical Pain: a Multicenter Real-World Study in China
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: GDKH001
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: The compound methyl salicylate liniment — The compound methyl salicylate liniment (Ammeltz) has been developed by Japan Sendai Kobayashi Pharmaceutical Co. and has been listed in Japan for many years. It is composed of various components, such as methyl salicylate, menthol, camphor, chlorpheniramine maleate, and thymol.
  Other Names: Ammeltz

SUMMARY:
The purpose of this phase Ⅳ clinical trial was to evaluate the safety and efficacy of compound methyl salicylate liniment (Ammeltz) in a real-life environment in China. This multicenter clinical trial was conducted at 22 hospitals/centers in China between May 2014 and March 2015.

The primary aim of the trial was to evaluate the safety of Ammeltz in a real-life environment. The secondary monitoring objective was to evaluate the efficacy of Ammeltz in the treatment of soft tissue injury pain in a real-life environment.

In principle, according to the guide for drug monitoring in production enterprises in China, the number of patients included in the statistical analysis of key drug monitoring should not be less than 3000 in order to provide ample information about the trial drug. Therefore, the sample size of this study was chosen to be 3600 cases, considering the dropout rate of the subjects.

DETAILED DESCRIPTION:
The investigators collected demographic data, vital signs, current medical history (type of soft tissue damage), and allergy history of the eligible patients on the day of Ammeltz prescription. At the same time, a doctor conducted the physical examination and evaluated the visual analog scale (VAS) score of each patient. On the seventh day of the drug administration (one course of the treatment lasts seven days), the investigator asked each patient by telephone about the actual use of the study drug, whether adverse events occurred, and about the self-assessment pain VAS score. On the 37th day of the treatment, the patients were interviewed again by telephone to inquire about the occurrence of adverse events .

The inclusion criteria for the patients were as follows: 1) age 3-75 years, male or female sex; 2) soft tissue pain caused by shoulder and neck pain, back pain, muscle pain, sprain, strain, contusion, muscle swelling and pain, and arthritis; local symptoms included pain, swelling, bruising, or tenderness; 3) signed informed consent and willing to participate in the study.

Patients were excluded if they met the following criteria: 1) allergy to any of the ingredients in this drug; 2) pregnant women, lactating women, and infants aged 0-3 years; 3) the affected area in the eye or mucous membranes, eczema, macules, wounds, and damaged skin; 4) patients without indications for the use of this drug.

ELIGIBILITY:
The inclusion criteria for the patients were as follows: 1) age 3-75 years, male or female sex; 2) soft tissue pain caused by shoulder and neck pain, back pain, muscle pain, sprain, strain, contusion, muscle swelling and pain, and arthritis; local symptoms included pain, swelling, bruising, or tenderness; 3) signed informed consent and willing to participate in the study.

Patients were excluded if they met the following criteria: 1) allergy to any of the ingredients in this drug; 2) pregnant women, lactating women, and infants aged 0-3 years; 3) the affected area in the eye or mucous membranes, eczema, macules, wounds, and damaged skin; 4) patients without indications for the use of this drug.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: people with soft tissue pain caused by shoulder and neck pain, back pain, muscle pain, sprain, strain, contusion, muscle swelling and pain, and arthritis; local symptoms included pain, swelling, bruising, or tenderness
Sampling Method: Probability Sample
Enrollment: 3600 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The adverse events | between May 2014 and March 2015
  On the seventh and the 37th day of the drug administration (one course of the treatment lasts seven days), the investigator asked each patient by telephone whether adverse events occurred.

SECONDARY OUTCOMES:
the self-assessment pain by VAS score | between May 2014 and March 2015
  On the seventh and the 37th day of the drug administration (one course of the treatment lasts seven days), the investigator asked each patient by telephone about the self-assessment pain VAS score.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo J, Hu X, Wang J, Yu B, Li J, Chen J, Nie X, Zheng Z, Wang S, Qin Q. Safety and efficacy of compound methyl salicylate liniment for topical pain: A multicenter real-world study in China. Front Pharmacol. 2022 Oct 21;13:1015941. doi: 10.3389/fphar.2022.1015941. eCollection 2022. PMID 36339533